CLINICAL TRIAL: NCT00240747
Title: Open-label, Multiple-dose, Phase III Study of the Population Pharmacokinetics of I.V. Synercid in 75 Pediatric Patients
Status: Terminated | Phase: Phase 3 | Type: Interventional
Sponsor: Pfizer (Industry)
Collaborators: Aventis Pharmaceuticals (Industry)
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: RP59500V-324
Record Dates: First submitted 2005-10-14; First posted 2005-10-18 (Estimated); Last update posted 2012-05-25 (Estimated); Status verified 2012-05

CONDITIONS: Gram-Positive Bacterial Infections
MeSH Terms: conditions — Gram-Positive Bacterial Infections | interventions — quinupristin-dalfopristin

INTERVENTIONS:
Drug: Synercid

SUMMARY:
Open-label, multicenter, multiple-dose, study of population pharmacokinetics of I.V. Synercid (7.5 mg/kg every 8 hours) in 75 pediatric patients. The purpose is to assess the population pharmacokinetics of Synercid in pediatric patients and to collect additional safety and efficacy data in pediatric patients.

ELIGIBILITY:
Inclusion Criteria:

* Serious, suspected or documented gram-positive infection

Exclusion Criteria:

-

Ages: 27 Weeks to 16 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Dates: Start 2000-06; Study Completion 2005-01

PRIMARY OUTCOMES:
Population pharmacokinetics

SECONDARY OUTCOMES:
Safety
Efficacy

CONTACTS AND LOCATIONS:
Overall Officials: George Talbot, M.D., Study Director — Yale University
Locations (6):
- United States (6):
  - Children's Hospital, Oakland, California
  - Children's Hospital of Orange County, Orange, California
  - Duke University Medical Center, Durham, North Carolina
  - Children's Hospital, Cincinnati, Ohio
  - The Cleveland Clinic, Cleveland, Ohio
  - Children's Hospital at Saint Francis, Tulsa, Oklahoma